CLINICAL TRIAL: NCT02124096
Title: Zoonotic Influenza Infections of Swine Origin at Ohio Agricultural Fairs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914092; 14-I-N092
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06-17

CONDITIONS: Influenza
Keywords: Zoonotic; Influenza; Infections; Ohio; Fairs
MeSH Terms: conditions — Influenza, Human; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- The flu is a very infectious and contagious virus that affects both people and pigs. Studies show that pigs can be sources of the flu virus in humans. Researchers want to know more about how the flu is transmitted from animals to people. If they know more about it, they can find better ways to prevent the flu and treat people who get sick from it.

Objective:

- To discover if flu viruses can be found in people exposed to pigs at Ohio agricultural fairs.

Eligibility:

- Volunteers 8 years of age and older who exhibit pigs at Ohio agricultural fairs.

Design:

* Before or on the first day of the fair, participants will fill out a short demographic and medical history form. They will also complete a two-page symptom questionnaire. This is a form that asks them about any flu symptoms they might have.
* Participants will have a nasal swab performed. The inside of the participant s nose will be rubbed with a swab to collect nasal fluid.
* Researchers will see participants 2 days later and 4 days later. During these visits, participants will again fill out a symptom questionnaire and have a nasal swab.

DETAILED DESCRIPTION:
The bidirectional transmission of influenza A viruses between animals and humans are clearly an important part of the complex dynamics of influenza evolution, however a thorough understanding of this process remains a mystery. The role of swine in overall human influenza evolution is unclear, but a long history of the study of swine origin influenza has revealed that influenza evolves in swine populations both in North America and Europe.

In 2009, a pandemic occurred with the emergence of the H1N1 pandemic (pdm) virus which was found to have originated from both a North American and European swine lineage, again reinforcing how viruses evolving in swine can lead to important human pathogens. Interestingly this virus was transmitted back into swine and birds in North America. In 2011, an H3N2 swine origin influenza virus known as the H3N2v and containing the H1N1pdm matrix genomic segment was reported causing human infections in multiple parts of the US. In 2012, these cases increased, especially during the summer months. Since 2011, 321 confirmed cases have been reported from 13 states including 107 cases in Ohio. Almost all of these cases have been linked to swine exposure on farms or at agricultural fairs.

Study of these zoonotic transmission events at agricultural fairs are necessary in order to better understand how and why these events occur, how human pathogens emerge, and how to potentially prevent events from occurring. These events could lead to new pandemics and epidemics so their prevention is crucial. The goal of this study is to examine rates of bidirectional zoonotic transmission at Ohio agricultural fairs. Through collection of viruses and host samples, we hope to begin to answer questions regarding how viruses cross species barriers, adapt to new hosts, and how these events could impact overall influenza virus evolution.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Volunteers greater than or equal to 8 years of age
* Parental consent if a participant is less than 18 years of age
* Willing to have samples stored for future research
* Willingness to complete all study procedures
* Daily or nearly daily contact with swine during selected agricultural fairs

EXCLUSION CRITERIA:

Any medical condition or circumstance that may make it unsafe for the participant to have nasal swab performed.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2014-04-25; Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Identification of influenza A virus infections occurring due to swinevariant influenza | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Ohio State University, College of Veterinary Medicine, Columbus, Ohio, United States

REFERENCES:
- [Background] Webster RG. The importance of animal influenza for human disease. Vaccine. 2002 May 15;20 Suppl 2:S16-20. doi: 10.1016/s0264-410x(02)00123-8. PMID 12110250
- [Background] Reid AH, Taubenberger JK. The origin of the 1918 pandemic influenza virus: a continuing enigma. J Gen Virol. 2003 Sep;84(Pt 9):2285-2292. doi: 10.1099/vir.0.19302-0. PMID 12917448
- [Background] Gray GC, McCarthy T, Capuano AW, Setterquist SF, Olsen CW, Alavanja MC. Swine workers and swine influenza virus infections. Emerg Infect Dis. 2007 Dec;13(12):1871-8. doi: 10.3201/eid1312.061323. PMID 18258038